CLINICAL TRIAL: NCT04411979
Title: Cognitive Function and Energy Metabolites in Schizophrenia: the Effect of Wearable Device-assisted Walking
Brief Title: Effects of 12 Weeks Walking on Cognitive Function in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOST 107-2635-B-182A-002; 201702283A3C601 (Other: Chang Gung Memorial Hospital)
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2018-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment-as-usual (No Intervention)
- treatment-as-usual plus aerobic walking (Experimental)
  Interventions: Other: treatment-as-usual plus aerobic walking

INTERVENTIONS:
Other: treatment-as-usual plus aerobic walking — aerobic walking
  Arms: treatment-as-usual plus aerobic walking

SUMMARY:
This study is a 12-week randomized-controlled clinical trial. It will be planned to conduct in a total of 120 male and female subjects from the Department of Psychiatry at Kaohsiung Chang Gung Memorial Hospital. Eligible subjects will be psychiatric patients, aged between 20-65 years old, who have psychiatric diagnosis of schizophrenia and fulfill the inclusion and exclusion criteria. The intervention with aerobic walking programs will be initiated after randomization for patients who continue their usual treatment. Subjects will be enrolled for 12 weeks aerobic walking treatment and randomly assigned to (1) treatment-as-usual, (2) treatment-as-usual plus aerobic walking. We will measure the treatment response to clarify the effect of aerobic walking in patients with schizophrenia. This study is being performed to investigate the possibly beneficial effects of aerobic walking on cognitive function and energy metabolites in schizophrenia.

DETAILED DESCRIPTION:
This 12-week randomized-controlled clinical trial will be planned to conduct in a total of 120 male and female subjects from the Department of Psychiatry at Kaohsiung Chang Gung Memorial Hospital. Eligible subjects will be psychiatric patients, aged between 20-65 years old, who have psychiatric diagnosis of schizophrenia and fulfill the inclusion and exclusion criteria. The intervention with aerobic walking programs will be initiated after randomization for patients who continue their usual treatment. Subjects will be enrolled for 12 weeks aerobic walking treatment and randomly assigned to (1) treatment-as-usual, (2) treatment-as-usual plus aerobic walking. The wearable watch will be used during the participants join the walking programs. We will measure the treatment response to investigate the effect of aerobic walking in patients with schizophrenia. This study is being performed to investigate the possibly beneficial effects of aerobic walking on cognitive function in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been diagnosed of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition criteria (DSM-5) criteria
2. The patient has the ability to complete the written informed consent

Exclusion Criteria:

1. The patient has been diagnosed with organic mental disorders, intelligence disability, dementia, major depressive disorder, bipolar affective disorder, and alcohol or substance use disorder
2. The patient has major systemic physical diseases, including cardiovascular diseases, uncontrollable arrhythmia, renal diseases, liver diseases or thyroid diseases
3. The patient has certified as physical disability
4. The patient is pregnant or has genetic diseases or infectious conditions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
cognitive function change | week 12
  cognitive function change assessed by Brief Assessment of Cognition in Schizophrenia
treatment change assessed by serum levels of energy metabolites (e.g., β-hydroxybutyrate) | week 12
  change assessment

SECONDARY OUTCOMES:
treatment change assessed by the Positive and Negative Syndrome Scale | week 12
  minimum value 30, maximum value 210; higher scores mean a worse outcome
treatment change assessed by peripheral blood metabolic profiles (e.g., plasma cholesterol level) | week 12
  change assessment
treatment change assessed by metabolic profiles (e.g., body weight in kilograms) | week 6, week 12
  change assessment
treatment change assessed by serum levels of inflammatory cytokines (e.g., IL-8) | week 12
  change assessment
treatment change assessed by 6-minute walk test | week 12
  change assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chi Huang, MD, Principal Investigator — Department of Psychiatry, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Department of Psychiatry, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No